CLINICAL TRIAL: NCT05719870
Title: A Multidisciplinary Approach to Improve Adherence to Medical Recommendations in Older Adults at Hospital Discharge
Brief Title: A Multidisciplinary Approach to Improve Adherence to Medical Recommendations in Older Adults
Acronym: APPROACH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Collaborators: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 947/2021/SPER/AOUFe
Record Dates: First submitted 2022-11-02; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-06

CONDITIONS: Medication Adherence; Aging; Multidisciplinary Communication; Fall; Hospital Discharge
MeSH Terms: conditions — Medication Adherence | interventions — Training Support

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the intervention vs. control group. The intervention will include: first, educational training of patients/caregivers at hospital discharge by a multidisciplinary team; second, after hospital discharge, a phone recall on the prescribed therapies and a one-week phone consultant service managed by a geriatrician, supported by the multidisciplinary team, to address potential concerns on prescribed treatments. Control group will follow usual care.
  After 7 days medication adherence will be assessed for both study groups through structured phone interviews.
  Over 30 and 90 days from discharge, data on falls, rehospitalizations and vital status will be collected through hospital records.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients hospitalized in the Geriatric Unit aged 60 years or older, that living in the community setting and who will be discharged at home and with expected survival >7 days.
  Interventions: Behavioral: Educational training
- Control group (No Intervention): Patients hospitalized in the Geriatric Unit aged 60 years or older, that living in the community setting and who will be discharged at home and with expected survival >7 days.
  The control group will be discharged following standard care procedures, and will receive only appropriate corrections and clarifications in case mistakes in the comprehension of the medical recommendations.

INTERVENTIONS:
Behavioral: Educational training — The intervention will include: first, educational training of patients/caregivers at hospital discharge by a multidisciplinary team; second, after hospital discharge, a phone recall on the prescribed therapies and a one-week phone consultant service managed by a geriatrician, supported by the multidisciplinary team, to address potential concerns on prescribed treatments.
  Arms: Intervention group

SUMMARY:
Background and overall goal: Poor comprehension and medication adherence are common in older people, especially after hospitalizations, in case of changes or prescriptions of new therapeutic regimes. The aim of this project is to evaluate the effectiveness of a multidomain intervention with an integrated care approach, in improving medication adherence in older people after hospital discharge. A secondary aim is investigate the determinants of poor comprehension and medication adherence in such individuals.

Target population: The project will involve older patients hospitalized in a Geriatric Department and discharged at home, and (when present) their caregivers.

Methods and assessments: Upon hospital discharge, data from the comprehensive geriatric assessment and information on the present hospitalization and prescribed therapies will be collected for all participants. The comprehension of medical recommendations reported in the discharge summary will be evaluated for all patients/caregiver before and after the routine explanation by treating physicians. Participants will be then randomized in intervention vs. control group. The intervention will include: first, educational training of patients/caregivers at hospital discharge by a multidisciplinary team; second, after hospital discharge, a phone recall on the prescribed therapies and a one-week phone consultant service managed by a geriatrician, supported by the multidisciplinary team, to address potential concerns on prescribed treatments. Control group will follow usual care. After 7 days medication adherence will be assessed for both study groups through structured phone interviews. At 30 and 90 days from discharge, data on falls, rehospitalizations and vital status will be collected through hospital records.

DETAILED DESCRIPTION:
Background and overall goal: Poor comprehension and medication adherence are common in older people, especially after hospitalizations, in case of changes or prescriptions of new therapeutic regimes. The aim of this project is to evaluate the effectiveness of a multidomain intervention with an integrated care approach, in improving medication adherence in older people after hospital discharge. Moreover, a secondary aim is to investigate the determinants of poor comprehension and medication adherence in such individuals.

Target population: The project will involve older patients hospitalized in a Geriatric Department and discharged at home, and (when present) their caregivers.

Methods and assessments: Upon hospital discharge, data from the comprehensive geriatric assessment and information on the present hospitalization and prescribed therapies will be collected for all participants. The comprehension of medical recommendations reported in the discharge summary will be evaluated for all patients/caregiver before and after the routine explanation by treating physicians. Participants will be then randomized in intervention vs. control group. The intervention will include: first, educational training of patients/caregivers at hospital discharge by a multidisciplinary team; second, after hospital discharge, a phone recall on the prescribed therapies and a one-week phone consultant service managed by a geriatrician, supported by the multidisciplinary team, to address potential concerns on prescribed treatments. Control group will follow usual care. After 7, 30 and 90 days, data on medication adherence, falls, rehospitalizations and vital status will be assessed for both study groups through structured phone interviews and hospital records.

ELIGIBILITY:
For the enrolment of the study participants, we will regularly monitor ward admissions, and potential eligibility of the patients will be evaluated by using the following inclusion criteria:

* Patients hospitalized in the Geriatric Units of the Padua and Ferrara University Hospitals
* Age 60 years or older
* Patients living in the community setting and who will be discharged at home
* Expected survival >7 days

Exclusion criteria:

* Patients discharged in long-term care facilities or other acute or post-acute wards
* No consent to participate in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Comprehension of medical recommendation at hospital discharge | At baseline (corresponding to hospital discharge)
  number of mistakes in recalling the prescribed therapy
Adherence to medical recommendations given at hospital discharge | 7 days after hospital discharge
  number of discrepancies in taking the prescribed therapy
Adherence to the recommendations provided by the occupational therapist at hospital discharge | 7 days after hospital discharge
  number of days per week of recommendations' adherence

SECONDARY OUTCOMES:
Mortality | 7, 30 and 90 days after hospital discharge
  Assessment of vital status through hospital records and telephone interviews
Number of falls | 30 and 90 days after hospital discharge
  Evaluation through structured telephone interviews
Number of emergency department visits | 30 and 90 days after hospital discharge
  Evaluation through structured telephone interviews
Number of rehospitalizations | 30 and 90 days after hospital discharge
  Evaluation through structured telephone interviews

CONTACTS AND LOCATIONS:
Overall Officials: Cateriina Trevisan, MD, PhD, Principal Investigator — Università degli Studi di Ferrara
Locations (2):
- Italy (2):
  - Geriatric Unit of Ferrara Hospital, Ferrara
  - Geriatric Unit of the Padua Central Hospital, Padua

REFERENCES:
- [Derived] Zanforlini BM, Sambo S, Devita M, Cignarella A, Vezzali F, Sturani S, Grandieri A, Noale M, Siviero P, Limongi F, Volpato S, Sergi G, Trevisan C; APPROACH working group. A multidisciplinary approach to improve adherence to medical recommendations in older adults at hospital discharge: The APPROACH study protocol. PLoS One. 2024 Apr 30;19(4):e0297238. doi: 10.1371/journal.pone.0297238. eCollection 2024. PMID 38687693